CLINICAL TRIAL: NCT04149054
Title: Mobile Health App to Reduce Diabetes in Latina Women With Prior Gestational Diabetes
Brief Title: Mobile Health App to Reduce Diabetes in Latina Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Environment and Health Group, Inc. (Industry)
Responsible Party: Principal Investigator, Patricia Weitzman, Principal Investigator, Environment and Health Group, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R44 MD009454A; R44MD009454 (NIH)
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Mobile health app called "Hola Bebe" — For the pilot, all participants received a mobile app that contained 6 interactive audio/written modules in Spanish and English on the following topics: healthy eating; physical activity; portion control; eating healthy while eating out; eating out in Chinese, Italian, Mexican restaurants; and eating out in fast food restaurants. As noted above, the mobile app was customizable to include personalized activity reminders/notifications, and tailored action plans, along with videos for easy at-home exercises and user-friendly, easy-to-follow recipes.

SUMMARY:
The proposed project sought to develop a culturally- and individually-tailored, plain-language Spanish/English mobile phone intervention for Latinas with prior gestational diabetes (GDM). The intervention is based on earlier in-person to online modification of the CDC-funded Diabetes Prevention Program (DPP), for women with prior GDM led by co-investigator Dr. Ellen Seely of Brigham and Women's Hospital.

DETAILED DESCRIPTION:
The specific aims of the study were as follows:

Primary Aim 1: Develop a culturally-tailored mobile phone intervention for Latinas with prior GDM based on Brigham & Women's Hospital online DPP.

Primary Aim 2: Conduct a pilot trial of the intervention.

Primary Aim 3:Evaluate implementation feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Latina women
* ages 19-45
* with prior gestational diabetes by Carpenter and Coustan criteria
* within the past 5 year validated by medical record review
* own an Android or iOS smartphone.

Exclusion Criteria:

* Diagnosis of pre-pregnancy diabetes(type 1,2, or secondary diabetes)
* underlying disease that might interfere with participation in study (e.g.,significant gastrointestinal conditions)
* taking certain medications (e.g., glucocorticoids)
* pregnancy/undergoing infertility treatment.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The intervention exclusively targeted Latina women who had gestational diabetes in a prior pregnancy.
Enrollment: 18 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Sallis Self Efficacy for Healthy Eating Scale | eight weeks
  20 item survey that asks respondents to rate, on a 5-point scale, their confident motivating themselves to eat healthy on a regular basis for at least six months.
Sallis Self Efficacy for Physical Activity Scale | eight weeks
  12 item survey that asks respondents to rate, on a 5-point scale, their confidence at motivating themselves to exercise on a regular basis for at least six months.

SECONDARY OUTCOMES:
Body weight | eight weeks
  Body weight

CONTACTS AND LOCATIONS:
Locations (1):
- Environment and Health Group, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share study protocol, informed consent, and final report with other researchers.
Supporting Information: Study Protocol
Time Frame: 6 months post-study

REFERENCES:
- [Derived] Seely EW, Weitzman PF, Cortes D, Romero Vicente S, Levkoff SE. Development and Feasibility of an App to Decrease Risk Factors for Type 2 Diabetes in Hispanic Women With Recent Gestational Diabetes (Hola Bebe, Adios Diabetes): Pilot Pre-Post Study. JMIR Form Res. 2020 Dec 31;4(12):e19677. doi: 10.2196/19677. PMID 33382039